CLINICAL TRIAL: NCT03743506
Title: An Instrumented Wobble Board to Present the Distribution and Center of Pressure in Dynamic Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mogi das Cruzes (Other)
Responsible Party: Principal Investigator, Terigi Augusto Scardovelli, Principal Investigator, University of Mogi das Cruzes
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 78363617.7.0000.5497
Record Dates: First submitted 2018-11-13; First posted 2018-11-16 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Balancing Interference
Keywords: Wobble board; center of pressure; dynamic balance; force platform

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Volunteers without motor abnormalities. (Experimental): The test was performed in a single, 30-minute session. The test is divided into two phases, with feedback and no feedback from the system. The order of phases was randomized. In each phase the volunteer will remain balanced on the wobble board for 15 seconds under the conditions of the phase. This test is repeated 3 times with a 30 seconds rest between them, then the next phase is performed. With feedback the volunteer can observe the system responses. Without feedback the volunteer can not observe the response of the system.
  Interventions: Diagnostic Test: With feedback; Diagnostic Test: Without feedback

INTERVENTIONS:
Diagnostic Test: With feedback — To evaluate the displacement of the center of pressure on the disc during the equilibration with feedback.
Diagnostic Test: Without feedback — To evaluate the displacement of the center of pressure on the disc during the equilibration without feedback.

SUMMARY:
This study quantified the displacement of the center of pressure in the computer in real time and record this data for future analyzes

DETAILED DESCRIPTION:
The wobble board is an unstable equilibrium platform, constant training on this platform generates an improvement in balance and strengthens the muscles, it is ideal for rehabilitation exercises and balance conditioning. However, these platforms do not provide quantitative data on exercises performed on it. And the force platform that provide this quantitative data is static, offering no difficulty in maintaining balance. In this way, a sensor board wobble board was developed using a conventional wobble board with a plate attached to it, between the plate and the platform are eight strain gauges sensors that are activated according to the position of the force applied on the platform, the values of the sensors are collected by software that demonstrates the point of greatest pressure on the disk and its displacement during the exercises, with this data it is possible to determine the stability of the user and observe their behavior during the exercises.

ELIGIBILITY:
Inclusion Criteria:

* Absence of musculoskeletal alteration in the lower limbs;
* consent form signed by the volunteer;
* with preserved cognitive

Exclusion Criteria:

* Present some impairment of the skeletal muscles of the lower limbs;
* Present cognitive deficit.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-11-10 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Pressure center displacement speed | 15 minutes
  The velocity at which the center of pressure moves during the test, divided into two steps, with three repetitions at each step, with a rest of 30 seconds at each repetition, was measured. Unit of measure: Centimeters per second (cm / s).

SECONDARY OUTCOMES:
Longest distance between points on X and Y axis | 15 minutes
  It was measured at the greatest distance of the center of pressure displacement on the X and Y axis during the test, divided into two steps, with three repetitions at each stage, with a rest of 30 seconds at each repetition. Unit of measurement: Centimeters (cm).

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro P Silva, Ph.D, Principal Investigator — University of Mogi das Cruzes
Locations (1):
- Alessandro Pereira da Silva, Mogi das Cruzes, São Paulo, Brazil